CLINICAL TRIAL: NCT04467476
Title: Effects of tDCS on Mechanical Power of the Leg Extensor Muscles of Healthy Subjects
Brief Title: Effects of tDCS on Anaerobic Power of Lower Limb Muscles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Clinical Professor - Physical Therapy Department, Universidade Federal do Piauí
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and anaerobic power
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (anodal) (Active Comparator): tDCS: 20 minutes, 2mA, over the motor cortex representation of lower limbs.
  Interventions: Device: Transcranial direct current stimulation
- tDCS (sham) (Sham Comparator): tDCS: 20 minutes (but 30s ON), 2mA, over the motor cortex representation of lower limbs.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation (NIBS) technique that has been investigated for the management of various health conditions. However, its ergogenic effect still has controversial results.

SUMMARY:
Anaerobic power and capacity are essential in many human activities, especially during sports practice that demand a high strength and power of the limbs. Transcranial direct current stimulation is a noninvasive technique that can modulate motor brain areas involved in motor functions and has the potential to optimize muscle capacity. However, their effects on mechanical power are lacking.

This study aims to investigate the effects of transcranial direct current stimulation (tDCS) on mechanical power in healthy subjects.

DETAILED DESCRIPTION:
In this study, a randomized, crossover, double-blind, placebo-controlled experimental design will be used. The 50 participants will be randomized into two groups: (1) Anodal tDCS(real) and (2) Sham tDCS. A single session of anodal and sham tDCS will be performed on each task (pre and post-jump test).

All evaluations will be performed by a single researcher who, like the participants, will not know which stimulation group will be participating. Subjects who agree to the conditions and sign the consent form may participate in the study. Participants who meet the eligibility criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no complaints of pain or any kind of discomfort in the musculoskeletal system

Exclusion Criteria:

* Musculoskeletal or neurological disorder
* Under medication
* Previous treatment with tDCS

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Mean anaerobic power | Pre and Post-test (immediately after tDCS)
  Mean anaerobic power will be evaluated by assessing the ground reaction forces (GRF) and the number of jumps in each test by means of the kinetic analysis of the 60-second vertical jump test (Bosco's Test).

SECONDARY OUTCOMES:
Peak anaerobic power | Pre and Post-test (immediately after tDCS)
  Peak anaerobic power will be evaluated by assessing the ground reaction forces (GRF) and the number of jumps in each test by means of the kinetic analysis of the 60-second vertical jump test (Bosco's Test).
Fatigue index | Pre and Post-test (immediately after tDCS)
  Fatigue index will be evaluated by assessing the ground reaction forces (GRF) and the number of jumps in each test by means of the kinetic analysis of the 60-second vertical jump test (Bosco's Test).
  The fatigue index corresponds to the power reduction rate expressed as a percentage and reveals the degree of reduction in the ability to produce strength and maintain exercise.
Rating of perceived exertion | Post-test (immediately after tDCS)
  The subjective feeling of effort will be assessed by the Borg scale for perceived effort. This is a 15-point numerical scale that ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion."

CONTACTS AND LOCATIONS:
Overall Officials: Fuas A Hazime, PhD, Principal Investigator — Department of Physical Therapy. Federal University of Piaui
Locations (1):
- Department of Physical Therapy. Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: Undecided